CLINICAL TRIAL: NCT04580550
Title: Evaluation of Axial Length Changes Between Pre and Postoperative Measurements
Brief Title: Axial Length Variability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vienna Institute for Research in Ocular Surgery (Other)
Responsible Party: Principal Investigator, Prim. Prof. Dr. Oliver Findl, MBA, Head of Department of Ophthalmology, Professor, Principal Investigator, MBA, Vienna Institute for Research in Ocular Surgery
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Axial length variability
Record Dates: First submitted 2020-09-30; First posted 2020-10-08 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Cataract Senile

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Axial length variability (Other): Aim of this study is to evaluate the magnitude of changes in pre and postoperative measurements of AL.
  Interventions: Other: Axial length variability

INTERVENTIONS:
Other: Axial length variability — Biometry (axial length measurement)is performed using the IOL Master 700 (Carl Zeiss Meditec AG, Jena, Germany) and Heidelberg Anterion (Heidelberg Engineering, Germany) pre and postoperatively.

SUMMARY:
The accuracy of IOL calculation relies on the one hand on axial length measurements and on the other hand on corneal and lens thickness measurements.

AL difference in pre and postoperative measurements may be caused by changes of lens parameters.

Aim of this study is to evaluate the magnitude of changes in pre and postoperative measurements of AL.

DETAILED DESCRIPTION:
This is a prospective observational, controlled and unmasked study that would include patients which undergo cataract presurgical examination, after patient signed written informed consent. For each patient only one eye will be included.

In total 50 eyes of 50 patients will be include. Due to missing previous data, the sample size is an approximation.

Prior to surgery, slit lamp examination and cataract grading (LOCS) is performed. Routine biometry is performed using the IOL Master 700 (Carl Zeiss Meditec AG, Jena, Germany) and Heidelberg Anterion (Heidelberg Engineering, Germany) for AL and lens measurement.

Additionally, evaluation of tilt and decentration will be performed using Purkinje meter device.

Follow-up examination will be performed three months after surgery and will contain: AL and lens measurement using the two ss-OCT biometery devices, lens evaluation (tilt and decentration of the IOL) using the Purkinje meter. Refractive outcome will be evaluated by determining best-corrected visual acuity and subjective refraction.

In women of childbearing age, a pregnancy test will be performed before inclusion into the study.

Main outcome variable:

• Extend of AL difference between pre- and postoperative measurements in both devices

Additional outcome variables:

* Agreement between the two ss-OCT devices in AL measurement
* Evaluation of lens parameter in AL differences between pre- and postoperative measurements
* Limit of agreement in lens tilt and decentration using two ss-OCT devices and Purkinje meter

ELIGIBILITY:
Inclusion Criteria:

* Uneventful cataract surgery
* Age 21 and older
* Axial length 24.00 mm and bigger
* CT Asphina 409 M lens implanted

Exclusion Criteria:

* Intra- or postoperative complication
* Relevant other ophthalmic diseases that are likely to influence the measurement outcome (as: with severe corneal pathology, severe macular degeneration, severe diabetic retinopathy, dens cataract, PEX syndrome, previous ocular surgery or trauma)
* Pregnancy

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Axial length variability | 3 months
  Evaluation of changes in axial length pre and post cataract surgery using two ss-OCT biometers

SECONDARY OUTCOMES:
Lens tilt and decentration | 3 months
  Evaluation of lens tilt and decantation using the Purkinje meter and two ss-OCT devices

CONTACTS AND LOCATIONS:
Locations (1):
- Hanusch Hospital, Ophthalmology department, Vienna, Austria